CLINICAL TRIAL: NCT00001246
Title: Brain Imaging of Childhood Onset Psychiatric Disorders, Endocrine Disorders and Healthy Volunteers
Status: Recruiting | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 890006; 89-M-0006
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01-09

CONDITIONS: Attention Deficit Hyperactivity Disorder; Schizophrenia; Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Hyperactivity Disorder; Twin; Sydenham's Chorea; Genetics; Development; Natural History
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Schizophrenia; Chorea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Our studies include data from typically developing youth, and individuals with a range of psychiatric presentations from behaviorally-defined (e.g. Childhood-Onset Schizophrenia, Autism Spectrum Disorder) as well as genetically-defined (e.g. Sex Chromosome Aneuploidy) groups. Participants span a wide age range (from 3 years of age upwards).

SUMMARY:
Magnetic Resonance Imaging (MRI) unlike X-rays and CT-scans does not use radiation to create a picture. MRI use as the name implies, magnetism to create pictures with excellent anatomical resolution. Functional MRIs are diagnostic tests that allow doctors to not only view anatomy, but physiology and function. It is for these reasons that MRIs are excellent methods for studying the brain.

In this study, researchers will use MRI to assess brain anatomy and function in X and Y chromosome variation, healthy volunteers, and patients with a variety of childhood onset psychiatric disorders. The disorders include attention deficit disorder, autism, congenital adrenal hyperplasia, childhood-onset schizophrenia, dyslexia, obsessive compulsive disorder, Sydenham's chorea, and Tourette's syndrome.

Results of the MRIs showing the anatomy of the brain and brain function will be compared across age, sex (gender), and diagnostic groups. Correlations between brain and behavioral measures will be examined for normal and clinical populations....

DETAILED DESCRIPTION:
Study Description:

This natural history protocol will have participants come to the NIH for brain imaging, psychological/psychiatric testing, and genetic characterization. Our core hypotheses are that many of the most severe neuropsychiatric disorders of childhood onset are associated with deviations from the path of normal brain development, the neuroanatomical substrates of which can be detected by magnetic resonance imaging.

Objectives:

Primary Objectives:

The long-term objectives of the protocol are to (1) map the neuroanatomic and neurophysiological trajectories of brain development; and (2) discern the influences, for good or ill, on those trajectories from demographic clinical, genetic, and environmental factors. Approximately half of the participants in our sample are typically developing. Clinical populations in our sample include participants with a variety of brain-based disorders, such as Autism, Attention-Deficit/Hyperactivity Disorder, Childhood Onset Schizophrenia, Dyslexia, Sydenham s Chorea, and Tourette s Syndrome.

Secondary Objectives:

To characterize the relationships among measures of behavior and cognition as well as amongst multimodal measures of brain organization.

Endpoints:

Primary Endpoint:

T1-weighted structural neuroimaging data which enable us to characterize how a range of anatomical brain phenotypes vary as a function of age, sex, behavioral/cognitive traits, diagnostic status and genotype.

Secondary Endpoints:

Data analyses also consider how these factors relate to other outcomes of interest including; gene expression levels, functional metrics from in vivo neuroimaging, and questionnaire/interview-based assessment of clinical features.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

Inclusion criteria for healthy controls

Participants consenting to participation in the study

-Over 3 years of age with no upper limit for age at time of enrollment.

Inclusion criteria for MRI scanner calibration project:

Participants will meet protocol criteria for adult healthy volunteers.

Inclusion criteria for affected participant populations:

-Male and female participants over 3 years of age with no upper limit for age (with the exception of the Down syndrome group - see below). Currently meet criteria for at least one of the following:

* DSM-IV (or other approved) criteria for one of the following clinical diagnoses: Obsessive Compulsive Disorder, Childhood Onset Schizophrenia, Turner Syndrome, Autism Spectrum Disorder, Asperger Syndrome, High Functioning Autism, Pervasive Development Disorder
* ICD-10 criteria for Congenital Adrenal Hyperplasia, Cushings Syndrome, Kallmann Syndrome, Androgen Insensitivity Syndrome.
* ADHD
* Chromosomal aneuploidies including Down s Syndrome and Sex chromosome aneuploidy as determined by karyotype (including XXX, XXXX, XXXXX, XXY, XXYY, XXXY, XXXXY, XYY, and XO).

Additional Inclusion criteria for Down Syndrome participants:

* Confirmed chromosomal diagnosis of Down syndrome.
* Age at entry into the study is 30 years or under. This upper age limit at study entry is being implemented for the Down syndrome group for several reasons. First, much of the research using magnetic resonance imaging with this population is focused on (older) adult populations and in particular the transition to early onset Alzheimer s disease. Because most (if not all) individuals with Down syndrome demonstrate some brain pathology consistent with Alzheimer s disease by age 30 (e.g., plaques and tangles; Mann & Esiri, 1989), we would like to enroll participants who are 30 years of age and under. Second, studying children and young adults with Down syndrome fills a significant gap in the literature, as there are very few structural magnetic resonance imaging studies of children and young adults with Down syndrome reported in the literature to date, and the majority of these studies are characterized by small samples of convenience (i.e., clinic populations). Thus, there is still a need to describe the developmental course of this disorder from early childhood to young adulthood. Such developmental research may help shed light on the causes of intellectual disability in Down syndrome and also identify individuals with the syndrome who are most at risk for experiencing the cognitive decline that is reported in the literature for some individuals after the age of 30 (Oliver et al., 1998).

Inclusion criteria for parents and siblings of affected participant populations:

Participants consenting to participation in the study

* Over 3 years of age with no upper limit for age at time of enrollment.
* Parents must have the ability to understand and provide informed consent to the study.

EXCLUSION CRITERIA:

NIMH staff and their immediate family are excluded from participation.

Exclusion criteria for healthy controls:

* Presence of severe psychiatric disorder (as diagnosed prior to participant study enrollment) in the participant. For these purposes, exclusionary severe psychiatric disorder includes schizophrenia and bipolar affective disorder.
* Presence or history of medical conditions known to affect cerebral anatomy.
* Dental braces.
* Contraindications for MRI scanning according to the NMR Center MRI Safety Screening Questionnaire and guidelines.
* For females who have reached menarche: Pregnancy or inability or unwillingness to undergo pregnancy testing.

Exclusion criteria for all affected participant populations, including parents and siblings of the affected participants:

* Dental braces.
* Contraindications for MRI scanning according to the NMR Center MRI Safety Screening Questionnaire and guidelines.
* For females who have reached menarche: Pregnancy or inability or unwillingness to undergo pregnancy testing.
* Evidence of another medical condition or traumatic event known to affect cerebral anatomy.
* A known genetic disorder (other than the condition under investigation) that would be expected to significantly impact findings from cognitive testing and/or neuroimaging.

Ages: 3 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Our studies include data from typically developing youth, and individuals with a range of psychiatric presentations from behaviorally-defined (e.g. Childhood-Onset Schizophrenia, Autism Spectrum Disorder) as well as genetically-defined (e.g. Sex Chromosome Aneuploidy) groups. Participants span a wide age range (from 3 years of age upwards).
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 1990-06-19 (Actual)

PRIMARY OUTCOMES:
Volumetric MRI Data | Ongoing
  Volumetric MRI Data

SECONDARY OUTCOMES:
Cognitive data | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Armin Raznahan, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share human data generated in this research for future research as follows@@@-Coded, linked data in an NIH-funded or approved public repository.@@@-Coded, linked data with approved outside collaborators under appropriate agreements.@@@@@@How and where will the data be shared?@@@@@@Data will be shared through:@@@-An NIH-funded or approved public repository: clinicaltrials.gov and dbGaP.@@@@@@-Approved outside collaborators under appropriate individual agreements.@@@@@@-Publication and/or public presentations.
Supporting Information: Study Protocol
Time Frame: When will the data be shared?@@@@@@-Within 1 year of completion of the primary endpoint.
Access Criteria: B. Data (including genomic data) and sample sharing plan@@@@@@Human Data Sharing Plan: This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals. Data from this study may be requested from other researchers 5 years after the completion of the primary endpoint by contacting Dr. Raznahan. Samples and data (including genomic data) will be shared with The University of Colorado.@@@@@@Data and samples may also be shared with approved collaborating laboratories at NIH or outside of NIH and/or submitted to NIH-designated repositories and databases if consent for sharing was obtained in the original consent form.

REFERENCES:
- [Derived] Hanson C, Blumenthal J, Clasen L, Guma E, Raznahan A. Influences of sex chromosome aneuploidy on height, weight, and body mass index in human childhood and adolescence. Am J Med Genet A. 2024 Feb;194(2):150-159. doi: 10.1002/ajmg.a.63398. Epub 2023 Sep 28. PMID 37768018
- [Derived] Liu S, Akula N, Reardon PK, Russ J, Torres E, Clasen LS, Blumenthal J, Lalonde F, McMahon FJ, Szele F, Disteche CM, Cader MZ, Raznahan A. Aneuploidy effects on human gene expression across three cell types. Proc Natl Acad Sci U S A. 2023 May 23;120(21):e2218478120. doi: 10.1073/pnas.2218478120. Epub 2023 May 16. PMID 37192167
- [Derived] Raznahan A, Rau S, Schaffer L, Liu S, Fish AM, Mankiw C, Xenophontos A, Clasen LS, Joseph L, Thurm A, Blumenthal JD, Bassett DS, Torres EN. Deep phenotypic analysis of psychiatric features in genetically defined cohorts: application to XYY syndrome. J Neurodev Disord. 2023 Feb 20;15(1):8. doi: 10.1186/s11689-023-09476-y. PMID 36803654
- [Derived] Guma E, Beauchamp A, Liu S, Levitis E, Clasen LS, Torres E, Blumenthal J, Lalonde F, Qiu LR, Hrncir H, MacKenzie-Graham A, Yang X, Arnold AP, Lerch JP, Raznahan A. A Cross-Species Neuroimaging Study of Sex Chromosome Dosage Effects on Human and Mouse Brain Anatomy. J Neurosci. 2023 Feb 22;43(8):1321-1333. doi: 10.1523/JNEUROSCI.1761-22.2022. Epub 2023 Jan 11. PMID 36631267
- [Derived] Csumitta KD, Gotts SJ, Clasen LS, Martin A, Raitano Lee N. Youth with Down syndrome display widespread increased functional connectivity during rest. Sci Rep. 2022 Jun 14;12(1):9836. doi: 10.1038/s41598-022-13437-1. PMID 35701489
- [Derived] Lee NR, Niu X, Zhang F, Clasen LS, Kozel BA, Smith ACM, Wallace GL, Raznahan A. Variegation of autism related traits across seven neurogenetic disorders. Transl Psychiatry. 2022 Apr 7;12(1):149. doi: 10.1038/s41398-022-01895-0. PMID 35393403
- [Derived] Mankiw C, Whitman ET, Torres E, Lalonde F, Clasen LS, Blumenthal JD, Chakravarty MM, Raznahan A. Sex-specific associations between subcortical morphometry in childhood and adult alcohol consumption: A 17-year follow-up study. Neuroimage Clin. 2021;31:102771. doi: 10.1016/j.nicl.2021.102771. Epub 2021 Jul 26. PMID 34359014
- [Derived] Warling A, Yavi M, Clasen LS, Blumenthal JD, Lalonde FM, Raznahan A, Liu S. Sex Chromosome Dosage Effects on White Matter Structure in the Human Brain. Cereb Cortex. 2021 Oct 22;31(12):5339-5353. doi: 10.1093/cercor/bhab162. PMID 34117759
- [Derived] Whitman ET, Liu S, Torres E, Warling A, Wilson K, Nadig A, McDermott C, Clasen LS, Blumenthal JD, Lalonde FM, Gotts SJ, Martin A, Raznahan A. Resting-State Functional Connectivity and Psychopathology in Klinefelter Syndrome (47, XXY). Cereb Cortex. 2021 Jul 29;31(9):4180-4190. doi: 10.1093/cercor/bhab077. PMID 34009243
- [Derived] Nadig A, Seidlitz J, McDermott CL, Liu S, Bethlehem R, Moore TM, Mallard TT, Clasen LS, Blumenthal JD, Lalonde F, Gur RC, Gur RE, Bullmore ET, Satterthwaite TD, Raznahan A. Morphological integration of the human brain across adolescence and adulthood. Proc Natl Acad Sci U S A. 2021 Apr 6;118(14):e2023860118. doi: 10.1073/pnas.2023860118. PMID 33811142
- [Derived] Wilson KE, Fish AM, Mankiw C, Xenophontos A, Warling A, Whitman E, Clasen L, Torres E, Blumenthal J, Raznahan A. Modeling familial predictors of proband outcomes in neurogenetic disorders: initial application in XYY syndrome. J Neurodev Disord. 2021 Mar 22;13(1):12. doi: 10.1186/s11689-021-09360-7. PMID 33752588
- [Derived] Raznahan A, Disteche CM. X-chromosome regulation and sex differences in brain anatomy. Neurosci Biobehav Rev. 2021 Jan;120:28-47. doi: 10.1016/j.neubiorev.2020.10.024. Epub 2020 Nov 7. PMID 33171144
- [Derived] Schmitt JE, Raznahan A, Liu S, Neale MC. The Heritability of Cortical Folding: Evidence from the Human Connectome Project. Cereb Cortex. 2021 Jan 1;31(1):702-715. doi: 10.1093/cercor/bhaa254. PMID 32959043
- [Derived] Liu S, Seidlitz J, Blumenthal JD, Clasen LS, Raznahan A. Integrative structural, functional, and transcriptomic analyses of sex-biased brain organization in humans. Proc Natl Acad Sci U S A. 2020 Aug 4;117(31):18788-18798. doi: 10.1073/pnas.1919091117. Epub 2020 Jul 20. PMID 32690678
- [Derived] Raznahan A. Editorial: Do Different Neurogenetic Disorders Impart Different Profiles of Psychiatric Risk? J Am Acad Child Adolesc Psychiatry. 2020 Sep;59(9):1022-1024. doi: 10.1016/j.jaac.2020.03.002. Epub 2020 Apr 12. PMID 32171632
- [Derived] Dworkin JD, Linn KA, Solomon AJ, Satterthwaite TD, Raznahan A, Bakshi R, Shinohara RT. A local group differences test for subject-level multivariate density neuroimaging outcomes. Biostatistics. 2021 Jul 17;22(3):646-661. doi: 10.1093/biostatistics/kxz058. PMID 31875881
- [Derived] Xenophontos A, Seidlitz J, Liu S, Clasen LS, Blumenthal JD, Giedd JN, Alexander-Bloch A, Raznahan A. Altered Sex Chromosome Dosage Induces Coordinated Shifts in Cortical Anatomy and Anatomical Covariance. Cereb Cortex. 2020 Apr 14;30(4):2215-2228. doi: 10.1093/cercor/bhz235. PMID 31828307
- [Derived] Bedford SA, Park MTM, Devenyi GA, Tullo S, Germann J, Patel R, Anagnostou E, Baron-Cohen S, Bullmore ET, Chura LR, Craig MC, Ecker C, Floris DL, Holt RJ, Lenroot R, Lerch JP, Lombardo MV, Murphy DGM, Raznahan A, Ruigrok ANV, Smith E, Spencer MD, Suckling J, Taylor MJ, Thurm A; MRC AIMS Consortium; Lai MC, Chakravarty MM. Large-scale analyses of the relationship between sex, age and intelligence quotient heterogeneity and cortical morphometry in autism spectrum disorder. Mol Psychiatry. 2020 Mar;25(3):614-628. doi: 10.1038/s41380-019-0420-6. Epub 2019 Apr 26. PMID 31028290
- [Derived] Schmitt JE, Raznahan A, Clasen LS, Wallace GL, Pritikin JN, Lee NR, Giedd JN, Neale MC. The Dynamic Associations Between Cortical Thickness and General Intelligence are Genetically Mediated. Cereb Cortex. 2019 Dec 17;29(11):4743-4752. doi: 10.1093/cercor/bhz007. PMID 30715232
- [Derived] Nadig A, Reardon PK, Seidlitz J, McDermott CL, Blumenthal JD, Clasen LS, Lalonde F, Lerch JP, Chakravarty MM, Raznahan A. Carriage of Supernumerary Sex Chromosomes Decreases the Volume and Alters the Shape of Limbic Structures. eNeuro. 2018 Nov 29;5(5):ENEURO.0265-18.2018. doi: 10.1523/ENEURO.0265-18.2018. eCollection 2018 Sep-Oct. PMID 30713992
- [Derived] McDermott CL, Seidlitz J, Nadig A, Liu S, Clasen LS, Blumenthal JD, Reardon PK, Lalonde F, Greenstein D, Patel R, Chakravarty MM, Lerch JP, Raznahan A. Longitudinally Mapping Childhood Socioeconomic Status Associations with Cortical and Subcortical Morphology. J Neurosci. 2019 Feb 20;39(8):1365-1373. doi: 10.1523/JNEUROSCI.1808-18.2018. Epub 2018 Dec 26. PMID 30587541
- [Derived] Joseph L, Farmer C, Chlebowski C, Henry L, Fish A, Mankiw C, Xenophontos A, Clasen L, Sauls B, Seidlitz J, Blumenthal J, Torres E, Thurm A, Raznahan A. Characterization of autism spectrum disorder and neurodevelopmental profiles in youth with XYY syndrome. J Neurodev Disord. 2018 Oct 22;10(1):30. doi: 10.1186/s11689-018-9248-7. PMID 30348076
- [Derived] Hamner T, Udhnani MD, Osipowicz KZ, Lee NR. Pediatric Brain Development in Down Syndrome: A Field in Its Infancy. J Int Neuropsychol Soc. 2018 Oct;24(9):966-976. doi: 10.1017/S1355617718000206. Epub 2018 May 23. PMID 29789029
- [Derived] Lenroot RK, Blumenthal JD, Wallace GL, Clasen LS, Lee NR, Giedd JN. A case-control study of brain structure and behavioral characteristics in 47,XXX syndrome. Genes Brain Behav. 2014 Nov;13(8):841-9. doi: 10.1111/gbb.12180. Epub 2014 Oct 27. PMID 25287572
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1989-M-0006.html